CLINICAL TRIAL: NCT03349385
Title: Multicenter Registry of Secondary Revascularization
Brief Title: Registry of Secondary Revascularization
Acronym: REVASEC
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Laboratorios Farmacéuticos Rovi, S.A. (Unknown); S&H MEDICAL SCIENCE SERVICE, S.L. (Other)
Responsible Party: Principal Investigator, Pablo Salinas, MD, Hospital San Carlos, Madrid
Other Study IDs: ROV-EPI-2017-01
Record Dates: First submitted 2017-11-11; First posted 2017-11-21 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease Progression; Coronary Artery Disease of Significant Bypass Graft; Stent Stenosis; Stent Restenosis; Coronary Arteriosclerosis
Keywords: Secondary revascularization; Repeat revascularization; Coronary revascularization; Coronary artery bypass graft
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study will evaluate patients with, at least, one previous procedure of coronary revascularization (surgical, percutaneous or both), that are referred for a new, clinically indicated, diagnostic coronary angiography, to describe their clinical characteristics, management, and prognosis, and will propose a prognosis-oriented classification.

DETAILED DESCRIPTION:
Secondary or repeated revascularization refers to any repeated coronary intervention following an index coronary revascularization procedure, and represents a wide proportion of patients received in catheterization laboratories. These patients have an increased complexity and worse outcomes than patients without previous revascularization. Clinical investigation has focused in lesion-specific treatments when a single previous revascularization fails, but there is paucity of patient-level information including complex patients with multiple revascularizations. Other gaps in evidence addressed by this study are the absence of a a prognosis-oriented classification of previously revascularized patients and a clinical meaningful definition of revascularization failure. The registry as well intends to provide insights on how secondary revascularization decisions are taken and long term prognosis after secondary revascularization.

The registry of secondary revascularization (in Spanish: Registro multicéntrico de reVAscularización SECundaria, REVASEC) is a multicenter, prospective, observational cohort study that incudes consecutive patients with at least one previous coronary revascularization undergoing a clinically indicated diagnostic coronary angiography, in different Spanish hospitals. The aims are describing the incidence, clinical profile, therapeutic management and prognosis of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Previous successful coronary revascularization, either percutaneous or surgical, in at least one vessel with diameter ≥2 mm
* Previous successful coronary revascularization must have been successful in at least one vessel and the patient must have been discharged after the previous revascularization
* Clinically indicated diagnostic coronary angiography
* Provide written informed consent

Exclusion Criteria:

* Inability or refusal to provide written informed consent
* Patient included in any other clinical trial in which the revascularization device is blind to patient or investigator, or is not commercially available
* Insufficient data about previous revascularizations
* Previous revascularization only on vessels of less than 2 mm or which was not successful in any vessel
* Previous percutaneous revascularization with simple plain old balloon angioplasty
* Index coronary angiography indicated as scheduled repeated angiography, planned percutaneous coronary intervention, or pre-surgical angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with at least one previous coronary revascularization undergoing a clinically indicated diagnostic coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 869 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Patient-oriented composite endpoint | 1 year
  Composite endpoint including: all-cause death, any myocardial infarction or any new unplanned revascularization

SECONDARY OUTCOMES:
Rates of individual components of primary outcome | 1 to 5 years
  Rates of individual components of primary outcomes: all-cause death, myocardial infarction or new unplanned revascularization
Composite endpoint at 2 to 5 years | 2 to 5 years
  Composite endpoint including: all-cause death, any myocardial infarction or new unplanned revascularization
Rate of failure of previous revascularization | baseline (assessed at index catheterization)
  Rate of failure of previous revascularization using the classical definition: >50% stent restenosis or >50% stenosis in a surgical graft
Recurrent angina (CCS class, patients reported) | 1 to 5 years
  Describe the presence of recurrent angina (CCS class) and analyze its predictors
Feasibility of secondary revascularization | per protocol, 1 month after index catheterization
  Define the rates of successful and complete revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Salinas, MD, PhD, Principal Investigator — Hospital San Carlos, Madrid
Locations (1):
- Hospital Clinico San Carlos, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salinas P, Vilchez-Tschischke JP, Noriega F, Macaya F, Rosillo S, Garcia-Camarero T, de la Torre-Hernandez JM, de Tapia B, Jimenez-Kockar M, Regueiro A, Flores-Umanzor E, Garcia-Blas S, Gonzalez-D'Gregorio J, Gomez-Menchero AE, Diaz-Fernandez JF, Rondan J, Amat-Santos I, Ojeda S, Diez-Gil JL, de Miguel Castro A, Lozano Ruiz-Poveda F, Fernandez-Diaz JA, Manzano MC, Cruz-Gonzalez I, Pascual Tejerina V, Garcia Perez-Velasco J, Serra A, Poveda-Andres JL, Macaya C, Escaned J. Design and Rationale for a Real-World Prospective, Multicenter Registry of Myocardial Revascularization Failure and Secondary Revascularization: The REVASEC Study. Cardiovasc Revasc Med. 2022 Jul;40:50-56. doi: 10.1016/j.carrev.2021.11.015. Epub 2021 Nov 16. PMID 34857473
- [Background] Salinas P, Garcia-Camarero T, Jimenez-Kockar M, Regueiro A, Garcia-Blas S, Gomez-Menchero AE, Ojeda S, Vilchez-Tschischke JP, Amat-Santos I, Diez-Gil JL, Rondan J, Lozano Ruiz-Poveda F, de Miguel Castro A, Manzano MC, Pascual-Tejerina V, Cruz-Gonzalez I, Garcia Perez-Velasco J, Fernandez-Diaz JA, Escaned J; REVASEC working group (collaborators). Myocardial revascularization failure among patients requiring cardiac catheterization and secondary revascularization in contemporary clinical practice: Results of the REVASEC multicenter registry. Catheter Cardiovasc Interv. 2023 Oct;102(4):608-619. doi: 10.1002/ccd.30804. Epub 2023 Aug 15. PMID 37582340